CLINICAL TRIAL: NCT02871778
Title: A Phase 2a, 2-part,Randomized, Double-blind, Placebo-controlled, Incomplete Block Crossover Study to Evaluate the Safety and Efficacy of VX-371 Solution for Inhalation With and Without Oral Ivacaftor in Subjects With Primary Ciliary Dyskinesia
Brief Title: Clearing Lungs With ENaC Inhibition in Primary Ciliary Dyskinesia
Acronym: CLEAN-PCD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parion Sciences (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PS-G202; 2015-004917-26 (EudraCT Number)
Record Dates: First submitted 2016-08-12; First posted 2016-08-18 (Estimated); Results first posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders | interventions — Saline Solution, Hypertonic; Sodium Chloride; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A: VX-371 in Hypertonic Saline (HS), Then HS (Experimental): Participants received 85 microgram (mcg) VX-371 diluted in 3 milliliter (mL) 4.2 percent (%) HS twice daily through oral nebulized inhalation from Day 1 through Day 29 in treatment period 1 followed by a 28 day washout period (from Day 29 through Day 56) and then received 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (from Day 57 through Day 85) in treatment period 2.
  Interventions: Drug: Hypertonic Saline; Drug: VX-371 + HS
- Part A: HS, Then VX-371 in HS (Experimental): Participants received 3 mL 4.2% HS through oral nebulized inhalation twice daily from Day 1 through Day 29 in treatment period 1 followed by a 28 day washout period (from Day 29 through Day 56) and then received 85 mcg VX-371 diluted in 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (from Day 57 through Day 85) in treatment period 2.
  Interventions: Drug: Hypertonic Saline; Drug: VX-371 + HS
- Part A: VX-371, Then Placebo (Experimental): Participants received 85 mcg VX-371 diluted in 3 mL 0.17% Saline (placebo) through oral nebulized inhalation twice daily from Day 1 through Day 29 in treatment period 1 followed by a 28 day washout period (from Day 29 through Day 56) and then received 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (from Day 57 through Day 85) in treatment period 2.
  Interventions: Drug: VX-371; Drug: Placebo (0.17% saline)
- Part A: Placebo, Then VX-371 (Experimental): Participants received 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily from Day 1 through Day 29 in treatment period 1 followed by a 28 day washout period (from Day 29 through Day 56) and then received 85 mcg VX-371 diluted in 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (from Day 57 through Day 85) in treatment period 2.
  Interventions: Drug: VX-371; Drug: Placebo (0.17% saline)
- Part B: VX-371 in HS + Ivacaftor (Experimental): Participants who were on 85 mcg VX-371 diluted in 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (from Day 57 through Day 85) in treatment period 2 continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 through Day 113) in treatment period 3.
  Interventions: Drug: VX-371 + HS; Drug: Ivacaftor
- Part B: HS + Ivacaftor (Experimental): Participants who were on 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (from Day 57 through Day 85) in treatment period 2 continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 through Day 113) in treatment period 3.
  Interventions: Drug: Hypertonic Saline; Drug: Ivacaftor
- Part B: VX-371 + Ivacaftor (Experimental): Participants who were on 85 mcg VX-371 diluted in 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (from Day 57 through Day 85) in treatment period 2 continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 through Day 113) in treatment period 3.
  Interventions: Drug: VX-371; Drug: Ivacaftor
- Part B: Placebo + Ivacaftor (Placebo Comparator): Participants who were on 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (from Day 57 through Day 85) in treatment period 2 continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 through Day 113) in treatment period 3.
  Interventions: Drug: Placebo (0.17% saline); Drug: Ivacaftor

INTERVENTIONS:
Drug: VX-371
  Arms: Part A: Placebo, Then VX-371; Part A: VX-371, Then Placebo; Part B: VX-371 + Ivacaftor
Drug: Hypertonic Saline
  Arms: Part A: HS, Then VX-371 in HS; Part A: VX-371 in Hypertonic Saline (HS), Then HS; Part B: HS + Ivacaftor
Drug: Placebo (0.17% saline)
  Arms: Part A: Placebo, Then VX-371; Part A: VX-371, Then Placebo; Part B: Placebo + Ivacaftor
Drug: VX-371 + HS
  Arms: Part A: HS, Then VX-371 in HS; Part A: VX-371 in Hypertonic Saline (HS), Then HS; Part B: VX-371 in HS + Ivacaftor
Drug: Ivacaftor
  Arms: Part B: HS + Ivacaftor; Part B: Placebo + Ivacaftor; Part B: VX-371 + Ivacaftor; Part B: VX-371 in HS + Ivacaftor

SUMMARY:
To evaluate the safety and efficacy of treatment with VX-371 with and without ivacaftor, and the effect of VX-371 with and without ivacaftor on quality of life (QOL) in subjects with primary ciliary dyskinesia (PCD).

ELIGIBILITY:
Inclusion Criteria:

* The subject must have evidence supportive of a PCD diagnosis.
* Subjects with percent predicted FEV1 of ≥40 to <90 percentage points
* Non-smoker for at least 90 days prior to the Screening Visit and less than a 5 pack-year lifetime history of smoking
* Stable regimen of medications and chest physiotherapy for the 28 days prior to Day 1
* If currently using daily inhaled HS, must be able to discontinue its use for the duration of the study.
* If taking daily chronic or chronic cycling antibiotics, has been on a consistent regimen for at least 4 months prior to the Screening Visit.
* Clinically stable (as deemed by the investigator) for at least 14 days prior to the Screening Visit
* Female subjects of childbearing potential must have a negative serum pregnancy test at the Screening Visit. Subjects of childbearing potential and who are sexually active must meet the contraception requirements.

Exclusion Criteria:

* Diagnosis of CF based on results of sweat chloride or nasal potential difference (NPD) tests or presence of 2 CF-causing mutations in CFTR gene.
* History of any organ transplantation or lung resection or chest wall surgery.
* Significant congenital heart defects, other than a laterality defect, at the discretion of the investigator
* Diagnosis of Cri du chat syndrome (chromosome 5p deletion syndrome).
* Inability to withhold short-acting bronchodilator use for 4 hours prior to clinic visit and long-acting bronchodilator use the night before the first and last clinic visit of each treatment period.
* Use of diuretics (including amiloride) or renin-angiotensin antihypertensive drugs
* Symptoms of acute upper or lower respiratory tract infection, acute pulmonary exacerbation, or treatment or was treated with systemic antibiotics for ear or sinus disease within 28 days before Day 1 (topical otic antibiotics allowed).
* History of significant intolerance to inhaled HS
* Pregnant and/or nursing females
* Any clinically significant laboratory abnormalities
* History of chronic B. cepacia complex or M. abscessus or M. avium
* Surgery that required general anesthesia and hospitalization within 3 months of Day 1

Additional Exclusion Criteria for Part B:

* In addition to the exclusion criteria above, subjects who participate in Part B and meet any of the following exclusion criteria will not be eligible to continue into Part B
* Unable to swallow tablets.
* Concomitant use of strong or moderate inhibitors or inducers of cytochrome P450 (CYP) 3A, including consumption of certain herbal medications (e.g., St. John's Wort), and grapefruit/grapefruit juice.
* Known hypersensitivity to ivacaftor.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Donn, Study Chair — Parion Sciences
Locations (34):
- United States (21):
  - Birmingham, Alabama
  - Palo Alto, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - New York, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Seattle, Washington
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- Copenhagen, Denmark
- Germany (3):
  - Münster, North Rhine-Westphalia
  - Hanover
  - Heidelberg
- Pisa, Italy
- Netherlands (2):
  - Amsterdam
  - Rotterdam
- Rabka-Zdrój, Poland
- United Kingdom (3):
  - Cambridge
  - London
  - Southampton

REFERENCES:
- [Derived] Ringshausen FC, Shapiro AJ, Nielsen KG, Mazurek H, Pifferi M, Donn KH, van der Eerden MM, Loebinger MR, Zariwala MA, Leigh MW, Knowles MR, Ferkol TW; CLEAN-PCD investigators and study team. Safety and efficacy of the epithelial sodium channel blocker idrevloride in people with primary ciliary dyskinesia (CLEAN-PCD): a multinational, phase 2, randomised, double-blind, placebo-controlled crossover trial. Lancet Respir Med. 2024 Jan;12(1):21-33. doi: 10.1016/S2213-2600(23)00226-6. Epub 2023 Aug 31. PMID 37660715

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of Part A and Part B. Total of 123 participants were randomized to 1 of 4 sequences in Part A to receive study drug.
Period: Part A: Treatment Period 1
Arm/Group | Part A: VX-371 in Hypertonic Saline (HS), Then HS | Part A: HS, Then VX-371 in HS | Part A: VX-371, Then Placebo | Part A: Placebo, Then VX-371 | Part B: VX-371 in HS + Ivacaftor | Part B: HS + Ivacaftor | Part B: VX-371 + Ivacaftor | Part B: Placebo + Ivacaftor
Started | 43 | 41 | 21 | 18 | 0 | 0 | 0 | 0
Safety Analysis Set | 44 (1 participant was randomized to receive HS in Period 1, but instead received VX-371 in HS in Period 1.) | 40 | 21 | 18 | 0 | 0 | 0 | 0
Completed | 40 | 37 | 18 | 16 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of consent (not due to adverse event) | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Noncompliant with study drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other withdrawal criteria met | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Wrong drug shipment | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A: Treatment Period 2
Arm/Group | Part A: VX-371 in Hypertonic Saline (HS), Then HS | Part A: HS, Then VX-371 in HS | Part A: VX-371, Then Placebo | Part A: Placebo, Then VX-371 | Part B: VX-371 in HS + Ivacaftor | Part B: HS + Ivacaftor | Part B: VX-371 + Ivacaftor | Part B: Placebo + Ivacaftor
Started | 40 | 37 | 18 | 16 | 0 | 0 | 0 | 0
Safety Analysis Set | 40 | 37 | 18 | 16 | 0 | 0 | 0 | 0
Completed | 37 | 35 | 17 | 15 | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Non-Compliant with Study Drug | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part B: Treatment Period 3
Arm/Group | Part A: VX-371 in Hypertonic Saline (HS), Then HS | Part A: HS, Then VX-371 in HS | Part A: VX-371, Then Placebo | Part A: Placebo, Then VX-371 | Part B: VX-371 in HS + Ivacaftor | Part B: HS + Ivacaftor | Part B: VX-371 + Ivacaftor | Part B: Placebo + Ivacaftor
Started | 0 | 0 | 0 | 0 | 11 (Out of 35 participants who were on VX-371 in HS in Treatment period 2 and completed Part A, 11 participants rolled-over to Part B.) | 27 (Out of 37 participants who were on HS in Treatment period 2 and completed Part A, 27 participants rolled-over to Part B.) | 7 (Out of 15 participants who were on VX-371 in Treatment period 2 and completed Part A, 7 participants rolled-over to Part B.) | 12 (Out of 17 participants who were on Placebo in Treatment period 2 and completed Part A, 12 participants rolled-over to Part B.)
Safety Analysis Set | 0 | 0 | 0 | 0 | 11 | 27 | 7 | 12
Completed | 0 | 0 | 0 | 0 | 10 | 26 | 6 | 12
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Part A Full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug in Part A and had a confirmed diagnosis of primary ciliary dyskinesia (PCD).
Groups:
- Part A: VX-371 in HS, Then HS: Participants received 85 mcg VX-371 diluted in 3 mL 4.2% HS twice daily through oral nebulized inhalation from Day 1 through Day 29 in treatment period 1 followed by a 28 day washout period (from Day 29 through Day 56) and then received 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (from Day 57 through Day 85) in treatment period 2.
- Total: Total of all reporting groups
Arm/Group | Part A: VX-371 in HS, Then HS | Part A: HS, Then VX-371 in HS | Part A: VX-371, Then Placebo | Part A: Placebo, Then VX-371 | Total
Number analyzed (Participants) | 43 | 41 | 21 | 18 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.19 (10.861) | 27.98 (13.104) | 27.62 (16.633) | 24.33 (12.866) | 27.80 (12.954)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 15 | 10 | 78
  Male | 14 | 17 | 6 | 8 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 0 | 7
  Not Hispanic or Latino | 41 | 37 | 18 | 18 | 114
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 1 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 1 | 5
  White | 39 | 36 | 17 | 14 | 106
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs included abnormal clinically significant findings for spirometry, clinical laboratory parameters, standard 12-lead electrocardiograms (ECGs), vital signs and pulse oximetry examinations. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 84 days that were absent before treatment or that worsened relative to pretreatment state. TEAEs included both serious and non-serious TEAEs.
Time Frame: Part A: From first dose of study drug up 84 days
Population: Part A safety set included all participants who received at least 1 dose of study drug in Part A.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: VX-371 in HS: Participants received 85 mcg VX-371 diluted in 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days in either treatment period 1 or 2.
- Part A: HS: Participants received 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days in either treatment period 1 or 2.
- Part A: VX-371: Participants received 85 mcg VX-371 diluted in 3 mL 0.17% Saline (placebo) through oral nebulized inhalation twice daily for 28 days in either treatment period 1 or 2.
- Part A: Placebo: Participants received 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days in either treatment period 1 or 2.
Arm/Group | Part A: VX-371 in HS | Part A: HS | Part A: VX-371 | Part A: Placebo
Number analyzed (Participants) | 81 | 80 | 37 | 36
Participants
  Participants with TEAEs | 52 | 46 | 22 | 23
  Participants with Serious TEAEs | 1 | 1 | 1 | 1

2. Primary Outcome: Part B: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs included abnormal clinically significant findings for spirometry, clinical laboratory parameters, standard 12-lead electrocardiograms (ECGs), vital signs and pulse oximetry examinations. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. TEAEs included both serious and non-serious TEAEs.
Time Frame: Part B: Day 85 up to 28 days after last dose of study drug (56 days)
Population: Part B safety set included all participants who received at least 1 dose of ivacaftor in Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: VX-371 in HS + IVA: Participants who received 85 mcg VX-371 diluted in 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (from Day 57 to Day 85) in treatment period 2, continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 to Day 113) in treatment period 3 (Part B).
- Part B: HS + IVA: Participants who received 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (from Day 57 to Day 85) in treatment period 2 continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 to Day 113) in treatment period 3 (Part B).
- Part B: VX-371 + IVA: Participants who received 85 mcg VX-371 diluted in 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (from Day 57 to Day 85) in treatment period 2, continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 to Day 113) in treatment period 3 (Part B).
- Part B: Placebo + IVA: Participants who received 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (from Day 57 to Day 85) in treatment period 2, continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 to Day 113) in treatment period 3 (Part B).
Arm/Group | Part B: VX-371 in HS + IVA | Part B: HS + IVA | Part B: VX-371 + IVA | Part B: Placebo + IVA
Number analyzed (Participants) | 11 | 27 | 7 | 12
Participants
  Participants with TEAEs | 5 | 17 | 5 | 9
  Participants with Serious TEAEs | 0 | 0 | 1 | 0

3. Primary Outcome: Part A: Absolute Change From Study Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Day 29
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. The study baseline is defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of study drug in the study.
Time Frame: Part A: Study Baseline, Day 29 of each treatment period
Population: Part A FAS included all randomized participants who received at least 1 dose of study drug in Part A and had a confirmed diagnosis of PCD. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of predicted FEV1
Arm/Group | Part A: VX-371 in HS | Part A: HS | Part A: VX-371 | Part A: Placebo
Number analyzed (Participants) | 78 | 75 | 34 | 34
Percentage of predicted FEV1 | 0.989 (0.7097) | -0.531 (0.7202) | -0.491 (1.0736) | -1.329 (1.0730)
Statistical Analysis 1: Comparison: Part A: VX-371 in HS vs Part A: HS; Test type: Superiority; p = 0.0437, Mixed-effects Model; Least Square (LS) Mean difference = 1.519, 95% CI 2-sided [0.044 to 2.995]
Statistical Analysis 2: Comparison: Part A: HS vs Part A: VX-371; Test type: Superiority; p = 0.9755, Mixed-effects Model; LS Mean difference = 0.040, 95% CI 2-sided [-2.509 to 2.589]
Statistical Analysis 3: Comparison: Part A: VX-371 in HS vs Part A: Placebo; Test type: Superiority; p = 0.0731, Mixed-effects Model; LS Mean difference = 2.318, 95% CI 2-sided [-0.22 to 4.856]
Statistical Analysis 4: Comparison: Part A: HS vs Part A: Placebo; Test type: Superiority; p = 0.5373, Mixed-effects Model; LS Mean Difference = 0.799, 95% CI 2-sided [-1.751 to 3.348]
Statistical Analysis 5: Comparison: Part A: VX-371 vs Part A: Placebo; Test type: Superiority; p = 0.453, Mixed-effects Model; LS Mean difference = 0.838, 95% CI 2-sided [-1.368 to 3.045]

4. Primary Outcome: Part B: Absolute Change From Study Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Day 29
Description: as for outcome 3
Time Frame: Study Baseline, Day 29 of Part B
Population: Part B FAS included all participants who had a confirmed diagnosis of PCD and received at least 1 dose of ivacaftor in Part B. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of predicted FEV1
Groups:
- Part B: VX-371 in HS + Ivacaftor: Participants who received 85 mcg VX-371 diluted in 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (from Day 57 to Day 85) in treatment period 2, continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 to Day 113) in treatment period 3 (Part B).
- Part B: HS + Ivacaftor: Participants who received 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (from Day 57 to Day 85) in treatment period 2 continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 to Day 113) in treatment period 3 (Part B).
- Part B: VX-371 + Ivacaftor: Participants who received 85 mcg VX-371 diluted in 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (from Day 57 to Day 85) in treatment period 2, continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 to Day 113) in treatment period 3 (Part B).
- Part B: Placebo + Ivacaftor: Participants who received 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (from Day 57 to Day 85) in treatment period 2, continued their inhaled study drug regimen from Treatment Period 2 and also received ivacaftor 150 mg tablet twice daily for 28 days (from Day 85 to Day 113) in treatment period 3 (Part B).
Arm/Group | Part B: VX-371 in HS + Ivacaftor | Part B: HS + Ivacaftor | Part B: VX-371 + Ivacaftor | Part B: Placebo + Ivacaftor
Number analyzed (Participants) | 10 | 26 | 6 | 12
Percentage of predicted FEV1 | 4.721 (1.9314) | 1.722 (1.1976) | -0.592 (2.5011) | -0.965 (1.8388)

5. Primary Outcome: Part B: Absolute Change From Part B Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Day 29
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Part B baseline was defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of ivacaftor in Part B and after the last dose in Period 2.
Time Frame: Part B Baseline, Day 29 of Part B
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percentage of predicted FEV1
Arm/Group | Part B: VX-371 in HS + Ivacaftor | Part B: HS + Ivacaftor | Part B: VX-371 + Ivacaftor | Part B: Placebo + Ivacaftor
Number analyzed (Participants) | 10 | 26 | 6 | 12
Percentage of predicted FEV1 | 2.528 (1.8633) | 1.678 (1.1414) | -1.018 (2.3797) | -2.040 (1.7427)

6. Secondary Outcome: Part A: Change From Study Baseline in Quality of Life-Primary Ciliary Dyskinesia (QOL-PCD) (Adult Version) Lower Respiratory Symptoms Domain Score at Day 29
Description: QOL- PCD adult version has following 10 domains: lower respiratory symptoms, emotional functioning, treatment burden, role, social functioning, vitality, health perception, upper respiratory symptoms, physical functioning and hearing symptoms. The total numbers of items in the lower respiratory symptoms domain are 6 in the questionnaire for adults. All items are scored using a 4-point Likert scale. Scaled score calculated as: [Sum of scores - (n*1)] / [(n*4) - (n*1)]*100. Where 'n' is the number of questions in domain. The total score range is from 0-100, where higher score indicates greater improvement. Change from study baseline >0 indicated improvement. The study baseline is defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of study drug in the study.
Time Frame: Study Baseline, Day 29 of Part A
Population: Part A FAS included all randomized participants who received at least 1 dose of study drug in Part A and had a confirmed diagnosis of PCD. Here, "overall number of participants analyzed" signifies adult participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: VX-371 in HS | Part A: HS | Part A: VX-371 | Part A: Placebo
Number analyzed (Participants) | 46 | 45 | 17 | 15
score on a scale | 4.23 (18.076) | 3.58 (16.715) | 0.98 (12.915) | 7.04 (16.728)

7. Secondary Outcome: Part B: Change From Study Baseline in Quality of Life-Primary Ciliary Dyskinesia (QOL-PCD) (Adult Version) Lower Respiratory Symptoms Domain Score at Day 29
Description: as for outcome 6
Time Frame: Study Baseline, Day 29 of Part B
Population: Part B FAS included all participants who had a confirmed diagnosis of PCD and received at least 1 dose of ivacaftor in Part B. Here, "overall number of participants analyzed" signifies adult participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: VX-371 in HS + Ivacaftor | Part B: HS + Ivacaftor | Part B: VX-371 + Ivacaftor | Part B: Placebo + Ivacaftor
Number analyzed (Participants) | 6 | 16 | 3 | 6
score on a scale | 16.67 (14.487) | 1.39 (17.153) | 7.41 (3.208) | -5.56 (23.307)

8. Secondary Outcome: Part B: Change From Part B Baseline in Quality of Life-Primary Ciliary Dyskinesia (QOL-PCD) (Adult Version) Lower Respiratory Symptoms Domain Score at Day 29
Description: QOL- PCD adult version has following 10 domains: lower respiratory symptoms, emotional functioning, treatment burden, role, social functioning, vitality, health perception, upper respiratory symptoms, physical functioning and hearing symptoms. The total numbers of items in the lower respiratory symptoms domain are 6 in the questionnaire for adults. All items are scored using a 4-point Likert scale. Scaled score calculated as: [Sum of scores - (n*1)] / [(n*4) - (n*1)]*100. Where 'n' is the number of questions in domain. The total score range is from 0-100, where higher score indicates greater improvement. Change from Part B baseline >0 indicated improvement. Part B baseline was defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of ivacaftor in Part B and after the last dose in Period 2.
Time Frame: Part B Baseline, Day 29 of Part B
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: VX-371 in HS + Ivacaftor | Part B: HS + Ivacaftor | Part B: VX-371 + Ivacaftor | Part B: Placebo + Ivacaftor
Number analyzed (Participants) | 6 | 16 | 3 | 6
score on a scale | 11.11 (15.713) | 1.39 (19.928) | 5.56 (16.667) | -7.41 (10.344)

9. Secondary Outcome: Part A: Change From Study Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score for Participants Aged Greater Than or Equals to (>=) 16 Years at Day 29
Description: SGRQ measured health-related quality of life among participants with respiratory diseases. It is a 40 items questionnaire grouped into three domains (Symptoms, Activity, and Impacts). Total scores range from 0 to 100. Higher score reflected worse quality of life. The study baseline is defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of study drug in the study.
Time Frame: Study Baseline, Day 29 of Part A
Population: Part A FAS included all randomized participants who received at least 1 dose of study drug in Part A and had a confirmed diagnosis of PCD. Here, "overall number of participants analyzed" signifies participants >=16 years of age evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: VX-371 in HS | Part A: HS | Part A: VX-371 | Part A: Placebo
Number analyzed (Participants) | 63 | 62 | 28 | 25
score on a scale | -1.28 (8.452) | -2.17 (6.462) | 1.54 (8.576) | -1.52 (9.082)

10. Secondary Outcome: Part B: Change From Study Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score for Participants Aged >=16 Years at Day 29
Description: as for outcome 9
Time Frame: Study Baseline, Day 29 of Part B
Population: Part B FAS included all participants who had a confirmed diagnosis of PCD and received at least 1 dose of ivacaftor in Part B. Here, "overall number of participants analyzed" signifies participants >=16 years of age evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: VX-371 in HS + Ivacaftor | Part B: HS + Ivacaftor | Part B: VX-371 + Ivacaftor | Part B: Placebo + Ivacaftor
Number analyzed (Participants) | 6 | 25 | 5 | 8
score on a scale | -1.69 (7.442) | -6.87 (6.571) | 0.78 (5.879) | 4.52 (16.995)

11. Secondary Outcome: Part B: Change From Part B Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score for Participants Aged >=16 Years at Day 29
Description: SGRQ measured health-related quality of life among participants with respiratory diseases. It is a 40 items questionnaire grouped into three domains (Symptoms, Activity, and Impacts). Total scores range from 0 to 100. Higher score reflected worse quality of life. Part B baseline was defined as the most recent non-missing measurement (scheduled or unscheduled) collected before the first dose of ivacaftor in Part B and after the last dose in Period 2.
Time Frame: Part B Baseline, Day 29 of Part B
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: VX-371 in HS + Ivacaftor | Part B: HS + Ivacaftor | Part B: VX-371 + Ivacaftor | Part B: Placebo + Ivacaftor
Number analyzed (Participants) | 6 | 25 | 5 | 8
score on a scale | -3.90 (4.331) | -2.64 (6.575) | 0.97 (7.561) | 3.19 (11.649)

ADVERSE EVENTS:
Time Frame: Part A: From first dose of study drug up to 84 days; Part B: Day 85 up to 28 days after last dose of study drug (56 days)
Description: Part A safety set included all participants who received at least 1 dose of study drug in Part A. Part B safety set included all participants who received at least 1 dose of ivacaftor in Part B.
Arm/Group | Part A: VX-371 in HS | Part A: HS | Part A: VX-371 | Part A: Placebo | Part B: VX-371 in HS + Ivacaftor | Part B: HS + Ivacaftor | Part B: VX-371 + Ivacaftor | Part B: Placebo + Ivacaftor
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/80 | 0/37 | 0/36 | 0/11 | 0/27 | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/81 | 1/80 | 1/37 | 1/36 | 0/11 | 0/27 | 1/7 | 0/12
Other Adverse Events (participants affected / at risk) | 40/81 | 27/80 | 12/37 | 16/36 | 5/11 | 15/27 | 4/7 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: VX-371 in HS (N=81) | Part A: HS (N=80) | Part A: VX-371 (N=37) | Part A: Placebo (N=36) | Part B: VX-371 in HS + Ivacaftor (N=11) | Part B: HS + Ivacaftor (N=27) | Part B: VX-371 + Ivacaftor (N=7) | Part B: Placebo + Ivacaftor (N=12)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: VX-371 in HS (N=81) | Part A: HS (N=80) | Part A: VX-371 (N=37) | Part A: Placebo (N=36) | Part B: VX-371 in HS + Ivacaftor (N=11) | Part B: HS + Ivacaftor (N=27) | Part B: VX-371 + Ivacaftor (N=7) | Part B: Placebo + Ivacaftor (N=12)
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Haemophilus test positive (Investigations) | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Moraxella test positive (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Forced expiratory volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Streptococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 4 | 3 | 3 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 3 | 0 | 0 | 2 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 8 | 3 | 3 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 8 | 7 | 2 | 6 | 3 | 4 | 0 | 3
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 5 | 6 | 0 | 1 | 0 | 3 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 2 | 2 | 0 | 3 | 1 | 0
Fatigue (General disorders) | 2 | 4 | 2 | 2 | 2 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 0 | 3 | 0 | 3 | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/78/NCT02871778/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT02871778/SAP_001.pdf